CLINICAL TRIAL: NCT06914570
Title: Cardiac Implantable Electronic Device- Induced Remodelling of Tricuspid Valve and Right Chambers
Acronym: CIED-REMTRIC
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C407
Record Dates: First submitted 2025-03-06; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Pacing, Artificial; Tricuspid Valve Regurgitation, Non-rheumatic
Keywords: Cardiac Implantable Electrical Devices; Tricuspid regurgitation; Three-dimensional echocardiography; Right ventricular remodeling
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIED: Patients undergoing new implantation of a CIED Inclusion criteria
  * Age ≥ 18 years
  * Patient is able and willing to give informed consent in written form before the index procedure
  * Patient understands the purpose, the potential risks and the benefits of the study and is willing to participate in all parts of the follow-up
  * Patients undergoing any new CIED implantation with or without transvalvular lead
  * Sufficient imaging quality on transthoracic echocardiography to assess TR severity grade and morphology of right-sided heart chambers Exclusion criteria
  * Previous or present CIED
  * Life expectancy < 12 months due to non-cardiac condition
  * Tricuspid valve stenosis of any severity or severe TR planned for intervention (transcatheter, surgical) within the next 12 months
  * Previous tricuspid valve intervention (transcatheter, surgical)

SUMMARY:
This single-center longitudinal study aims to evaluate the occurrence and clinical impact of tricuspid regurgitation (TR) after cardiac-implanted-electronic-device (CIED) implantation by comprehensive echocardiographic assessment, including advanced three-dimensional (3D) transthoracic and transesophageal imaging.

The primary objective of this study is to assess the prevalence and leading mechanism of new or worsening TR, defined as an increase of at least one grade on a five-grade scale, after new CIED implantation.

Secondary objectives include clinical and echocardiographic endpoints at discharge, three months, one year, and annually for up to five years.

They can be summarized as follows:

1. to evaluate morphological and functional changes (remodeling) of the tricuspid valve (TV) apparatus and right-sided heart chambers in patients undergoing new CIED implantation.
2. to identify risk factors for new or worsening TR after CIED implantation on an anatomical, procedural, and clinical level.
3. to determine the clinical impact of new or worsening TR after CIED implantation.
4. to explore the treatment strategies for lead-related TR (observational).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient able and willing to give informed consent in written form before the index procedure
* Patient understands the purpose, the potential risks as well as benefits of the study and is willing to participate in all parts of the follow-up
* Patients undergoing any new CIED implantation with or without transvalvular lead
* Sufficient imaging quality on transthoracic echocardiography to assess TR severity grade and morphology of right-sided heart chambers

Exclusion Criteria:

* Previous or present CIED
* Life expectancy < 12 months due to non-cardiac condition
* Tricuspid valve stenosis of any severity or severe TR planned for intervention (transcatheter, surgical) within the next 12 months
* Previous tricuspid valve intervention (transcatheter, surgical)
* Participation in another study, which would lead to deviations from this trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing new implantation of a CIED
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-02-24 (Estimated)

PRIMARY OUTCOMES:
Change in TR at least one grade after new CIED implantation | 5 years
  TR severity grade assessed using echocardiographic multi-parametric approach, including 3D echocardiography if possible.

SECONDARY OUTCOMES:
Incidence of mortality (all-cause, cardiovascular, non-cardiovascular) | 5 years
Incidence of heart failure Hospitalization or any change in diuretic dosage or need for intravenous diuretics | 1 year, and annually through 5 years
New York Heart Association (NYHA) functional class | at 1 day, 3 months, 1 year, and annually through 5 years
Incidence of tricuspid valve intervention (either transcatheter or surgical) | 1 year, and annually through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Badano, MD, Ph.D., Principal Investigator — Istituto Auxologico Italiano, IRCCS
Locations (1):
- San Luca Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Depends on subscription of a Data transfer agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: Researchers who are members of Institutions who will subscribe a data transfer agreement for this specific study
URL: https://zenodo.org/

REFERENCES:
- [Background] Seo J, Kim DY, Cho I, Hong GR, Ha JW, Shim CY. Prevalence, predictors, and prognosis of tricuspid regurgitation following permanent pacemaker implantation. PLoS One. 2020 Jun 26;15(6):e0235230. doi: 10.1371/journal.pone.0235230. eCollection 2020. PMID 32589674
- [Background] Kanawati J, Ng ACC, Khan H, Yu C, Hyun K, Abed H, Kritharides L, Sy RW. Long-Term Follow-Up of Mortality and Heart Failure Hospitalisation in Patients With Intracardiac Device-Related Tricuspid Regurgitation. Heart Lung Circ. 2021 May;30(5):692-697. doi: 10.1016/j.hlc.2020.08.028. Epub 2020 Oct 31. PMID 33132050
- [Background] Papageorgiou N, Falconer D, Wyeth N, Lloyd G, Pellerin D, Speechly-Dick E, Segal OR, Lowe M, Rowland E, Lambiase PD, Chow AW, Bhattacharyya S. Effect of tricuspid regurgitation and right ventricular dysfunction on long-term mortality in patients undergoing cardiac devices implantation: >10-year follow-up study. Int J Cardiol. 2020 Nov 15;319:52-56. doi: 10.1016/j.ijcard.2020.05.062. Epub 2020 May 27. PMID 32470533
- [Background] Delling FN, Hassan ZK, Piatkowski G, Tsao CW, Rajabali A, Markson LJ, Zimetbaum PJ, Manning WJ, Chang JD, Mukamal KJ. Tricuspid Regurgitation and Mortality in Patients With Transvenous Permanent Pacemaker Leads. Am J Cardiol. 2016 Mar 15;117(6):988-92. doi: 10.1016/j.amjcard.2015.12.038. Epub 2016 Jan 6. PMID 26833208
- [Background] Al-Bawardy R, Krishnaswamy A, Rajeswaran J, Bhargava M, Wazni O, Wilkoff B, Tuzcu EM, Martin D, Thomas J, Blackstone E, Kapadia S. Tricuspid regurgitation and implantable devices. Pacing Clin Electrophysiol. 2015 Feb;38(2):259-66. doi: 10.1111/pace.12530. Epub 2014 Nov 7. PMID 25377489
- [Background] Hoke U, Auger D, Thijssen J, Wolterbeek R, van der Velde ET, Holman ER, Schalij MJ, Bax JJ, Delgado V, Marsan NA. Significant lead-induced tricuspid regurgitation is associated with poor prognosis at long-term follow-up. Heart. 2014 Jun;100(12):960-8. doi: 10.1136/heartjnl-2013-304673. Epub 2014 Jan 21. PMID 24449717
- [Background] Baquero GA, Yadav P, Skibba JB, Banchs JE, Linton-Frazier LN, Lengerich EJ, Samii SM, Penny-Peterson E, Wolbrette DL, Luck JC, Naccarelli GV, Gonzalez MD. Clinical significance of increased tricuspid valve incompetence following implantation of ventricular leads. J Interv Card Electrophysiol. 2013 Dec;38(3):197-202. doi: 10.1007/s10840-013-9826-2. PMID 24022757